CLINICAL TRIAL: NCT06312436
Title: The Effectiveness of Resuscitative Endovascular Balloon Occlusion of the Aorta (REBOA) for Trauma Patients With Uncontrolled Haemorrhage: Study Protocol for a Target Trial and Its Emulation
Brief Title: The AT-REBOA Target Trial
Acronym: AT-REBOA
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: AT-REBOA
Record Dates: First submitted 2024-02-27; First posted 2024-03-15 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Hemorrhage; Shock, Traumatic; Cardiac Arrest Due to Trauma; Polytrauma
MeSH Terms: conditions — Hemorrhage; Shock, Traumatic; Multiple Trauma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- REBOA group: After allocation, access to a femoral artery is swiftly established by either ultrasound-guided puncture or via surgical cut-down. In parallel major haemorrhage protocol transfusion and further diagnostics are being carried out. Balloon occlusion is then achieved by placing a balloon catheter (ER-REBOA catheter, Prytime Medical®, Boerne, TX, USA) into aortic zone I (supradiaphragmatic) or III (aortic bifurcation) according to clinician decision based on injury pattern. Continuing management, including further computed tomography diagnostics and damage control interventions (operative or angioembolisation) and ongoing transfusions are undertaken according to patient status.
  Interventions: Procedure: Resuscitative Endovascular Balloon Occlusion of the Aorta (REBOA)
- Control group: After allocation, major haemorrhage protocol transfusion and all resuscitative measures except REBOA are performed. Continuing management, including further computed tomography diagnostics and damage control interventions (operative or angioembolisation) and ongoing transfusions are undertaken according to patient status.

INTERVENTIONS:
Procedure: Resuscitative Endovascular Balloon Occlusion of the Aorta (REBOA) — Temporary aortic occlusion can limit haemorrhage, can help to maintain perfusion to the heart and brain, and may be associated with improved survival.
  Groups: REBOA group

SUMMARY:
Temporary aortic occlusion can limit haemorrhage, can help to maintain perfusion to the heart and brain, and may be associated with improved survival. Resuscitative Endovascular Balloon Occlusion of the Aorta (REBOA) potentially provides a relatively quick means of achieving this temporary control.

In the past years, studies have tried to evaluate the benefit for this method with conflicting results. The previous UK-REBOA trial has not found any benefit in the intervention group and has even hinted at possible harm caused by the intervention. A major limitation of this study is the low number of interventions performed in participating trauma centres and the associated potentially insufficient experience with REBOA.

The aim of this study is to evaluate the effectiveness of REBOA in a setting with already experienced providers.

ELIGIBILITY:
Inclusion criteria:

* aged, or believed to be aged, 16 years or above
* confirmed or suspected life-threatening torso or lower body trauma
* thought to benefit from trauma resuscitation with REBOA

Exclusion criteria:

* penetrating chest trauma
* known or suspected pregnancy at presentation
* prehospital thoracotomy
* severe burns injuries.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target trial seeks to enrol patients in the trauma room who are thought to be at imminent risk of dying from acute blood loss due to non-compressible torso or lower body haemorrhage.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
30-day in-hospital mortality | 30 days

SECONDARY OUTCOMES:
3-hour mortality | 3 hours
6-hour mortality | 6 hours
24-hour mortality | 24 hours
90-day mortality | 90 days
Intensive Care Unit length of stay | within 6 months
  days
Hospital length of stay | within 6 months
  days
Blood product use | 48 hours
  amount of packed red blood cells, amount of fresh frozen plasma, amount of thrombocyte concentrates
Use of whole body computed tomography | during resuscitation care phase within 3 hours
damage control procedure performed | during resuscitation phase within 3 hours
  operation or angioembolisation
Time to damage control procedure | during resuscitation phase within 3 hours
  operation or angioembolisation
Rate of complications | within 6 months
  acute kidney injury °III, use of renal replacement therapy, arterial thrombosis or embolism, limb ischaemia, vascular injury, compartment syndrome requiring fasciotomy
Cause of death | within 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- Austria (2):
  - University Medical Centre Graz, Graz, Styria
  - Center for Medical Data Science, Vienna

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stannard A, Eliason JL, Rasmussen TE. Resuscitative endovascular balloon occlusion of the aorta (REBOA) as an adjunct for hemorrhagic shock. J Trauma. 2011 Dec;71(6):1869-72. doi: 10.1097/TA.0b013e31823fe90c. No abstract available. PMID 22182896
- [Background] Jansen JO, Hudson J, Cochran C, MacLennan G, Lendrum R, Sadek S, Gillies K, Cotton S, Kennedy C, Boyers D, Ferry G, Lawrie L, Nath M, Wileman S, Forrest M, Brohi K, Harris T, Lecky F, Moran C, Morrison JJ, Norrie J, Paterson A, Tai N, Welch N, Campbell MK; UK-REBOA Study Group; Aylwin C, Bew D, Brooks A, Chinery J, Cowlam T, Frith D, George A, Hudson A, Johnstone P, Mahmood A, Novak A, O'Meara M, Reid S, Sattout A, Smith C, Stansfield T, Thompson J. Emergency Department Resuscitative Endovascular Balloon Occlusion of the Aorta in Trauma Patients With Exsanguinating Hemorrhage: The UK-REBOA Randomized Clinical Trial. JAMA. 2023 Nov 21;330(19):1862-1871. doi: 10.1001/jama.2023.20850. PMID 37824132
- [Derived] Hallmann B, Honnef G, Eibinger N, Eichlseder M, Posch M, Puchwein P, Zoidl P, Zajic P. Resuscitative endovascular balloon occlusion of the aorta for trauma patients with uncontrolled hemorrhage: a retrospective target trial emulation (the AT-REBOA target trial). Eur J Emerg Med. 2025 Jun 1;32(3):202-209. doi: 10.1097/MEJ.0000000000001183. Epub 2024 Sep 24. PMID 39745669